CLINICAL TRIAL: NCT04806503
Title: A Randomized, Placebo-controlled, Double-masked, Multi-center, Dose-ranging Study to Evaluate the Safety, and Efficacy of UNR844 in Subjects With Presbyopia
Brief Title: A Dose-ranging Study to Evaluate the Safety and Efficacy of UNR844 in Subjects With Presbyopia.
Acronym: READER
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was discontinued by the Sponsor because it did not achieve the primary objective.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CUNR844A2202
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Presbyopia
Keywords: loss of elasticity in lens; lens; lens disorder; loss of near vision; Presbyopia; UNR844; farsightedness
MeSH Terms: conditions — Presbyopia; Lens Diseases; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- UNR844 5 mg/mL (Experimental): UNR844 5 mg/mL ophthalmic solution; one drop twice-a-day for three months
  Interventions: Drug: UNR844
- UNR844 13.3 mg/mL (Experimental): UNR844 13.3 mg/mL 1 ophthalmic solution; one drop twice-a-day for three months
  Interventions: Drug: UNR844
- UNR844 23 mg/mL (Experimental): UNR844 23 mg/mL ophthalmic solution; one drop twice-a-day for three months
  Interventions: Drug: UNR844
- UNR844 30 mg/mL (Experimental): UNR844 30 mg/mL ophthalmic solution; one drop twice-a-day for three months
  Interventions: Drug: UNR844
- Placebo Ophthalmic Solution (Placebo Comparator): placebo ophthalmic solution; one drop twice-a-day for three months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UNR844 — Ophthalmic solution for topical ocular administration
  Other Names: EV06
  Arms: UNR844 13.3 mg/mL; UNR844 23 mg/mL; UNR844 30 mg/mL; UNR844 5 mg/mL
Drug: Placebo — Placebo
  Other Names: Vehicle
  Arms: Placebo Ophthalmic Solution

SUMMARY:
Study of safety and efficacy of UNR844 in subjects with presbyopia.

DETAILED DESCRIPTION:
This was a randomized, placebo-controlled, double-masked,multi-arm, parallel-group, multi-center 13-month study which consisted of:

* A 1 week run-in period
* A 3-month treatment course with UNR844 and/or Placebo
* A 9-month treatment holiday period Participants were randomized equally to one of five treatment arms: UNR844 5 mg/mL,UNR844 13.3 mg/mL, UNR844 23 mg/mL, UNR844 30 mg/mL, or Placebo eye drops twice-a-day for three months.

Participants underwent a 1 week run-in period where they were assessed for entry criteria during the Screening visit. During the run-in period, participants self-administered 1 drop of artificial tears twice-a-day (1 drop in the morning and 1 drop in the evening) in each eye at home. This run-in period was designed to help minimize any potential variability in distance corrected near visual acuity (DCNVA) caused due to initial ocular surface issues and help to establish an accurate baseline prior to randomization. The run-in period was to help exclude participants with a change in DCNVA of 0.10 logMAR difference between Screening and Baseline.

This study was conducted to determine the optimum dose of UNR844 treatment and the duration of effect of UNR844 treatment for further development.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any assessment is performed
* Impaired near vision in each eye and when using both eyes, without any near correction
* Need a certain level of near correction

Exclusion Criteria:

* Impaired distance vision in either eye, with distance correction (if any)
* Severe short- or long-sightedness
* Any significant medical or clinical conditions affecting vision, the eyes or general health

Ages: 45 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 234 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- United States (11):
  - Novartis Investigative Site, Laguna Hills, California
  - Novartis Investigative Site, Newport Beach, California
  - Novartis Investigative Site, Largo, Florida
  - Novartis Investigative Site, Lake Villa, Illinois
  - Novartis Investigative Site, Pittsburg, Kansas
  - Novartis Investigative Site, Washington, Missouri
  - Novartis Investigative Site, Kingston, Pennsylvania
  - Novartis Investigative Site, Sioux Falls, South Dakota
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Smyrna, Tennessee
  - Novartis Investigative Site, San Antonio, Texas
- Australia (2):
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, East Melbourne, Victoria
- Canada (4):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Kitchener, Ontario
  - Novartis Investigative Site, Waterloo, Ontario
  - Novartis Investigative Site, Québec, Quebec
- Japan (2):
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shinjuku Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://clinicalstudydatarequest.com/

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1562

RESULTS

PARTICIPANT FLOW:
Groups:
- UNR844 13.3 mg/mL: UNR844 13.3 mg/mL ophthalmic solution; one drop twice-a-day for three months
Period: Overall Study
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Started | 48 | 48 | 44 | 48 | 46
Completed | 46 | 47 | 42 | 46 | 45
Not Completed | 2 | 1 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution | Total
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46 | 234
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (2.61) | 50.9 (2.80) | 51.0 (2.94) | 50.5 (2.66) | 51.2 (2.80) | 50.9 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 28 | 27 | 29 | 23 | 135
  Male | 20 | 20 | 17 | 19 | 23 | 99
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 11 | 9 | 10 | 11 | 11 | 52
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 2 | 2 | 1 | 14
  White | 32 | 34 | 32 | 34 | 34 | 166
  More than one race | 1 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Characterize Dose-response of UNR844 for Change From Baseline in Binocular Distance-corrected Near Visual Acuity (DCNVA) at Month 3
Description: Characterize dose response of UNR844 as measured by change from baseline at Month 3 in binocular DCNVA (without near correction) in Logarithm of Minimum Angle of Resolution (logMAR), at 40cm. A low logMAR score represents good vision while a high logMAR score represents bad vision.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
logMAR | -0.106 (0.0186) | -0.110 (0.0188) | -0.136 (0.0203) | -0.101 (0.0185) | -0.112 (0.0194)
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.817, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.006, 95% CI 2-sided [-0.045 to 0.056], Standard Error of Mean 0.0258
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.946, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.002, 95% CI 2-sided [-0.050 to 0.053], Standard Error of Mean 0.0262
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.380, Mixed-effect Model for Repeated Measures; Least Squares Mean = -0.024, 95% CI 2-sided [-0.077 to 0.029], Standard Error of Mean 0.0270
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.667, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.011, 95% CI 2-sided [-0.039 to 0.062], Standard Error of Mean 0.0258

2. Secondary Outcome: Characterize Dose Response of UNR844 as Measured by Change From Baseline in Monocular (Worse-seeing Eye) Distance-corrected Near Visual Acuity (DCNVA) at Month 3
Description: Characterize dose response of UNR844 as measured by change from baseline at Month 3 in monocular (worse-seeing eye) DCNVA in Logarithm of Minimum Angle of Resolution (logMAR), at 40 cm. A low logMAR score represents good vision while a high logMAR score represents bad vision.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
logMAR | -0.125 (0.0217) | -0.121 (0.0220) | -0.143 (0.0241) | -0.112 (0.0216) | -0.146 (0.0228)
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.474, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.022, 95% CI 2-sided [-0.038 to 0.081], Standard Error of Mean 0.0304
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.419, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.025, 95% CI 2-sided [-0.036 to 0.086], Standard Error of Mean 0.0309
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.914, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.003, 95% CI [-0.060 to 0.067], Standard Error of Mean 0.0322
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.263, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.034, 95% CI 2-sided [-0.026 to 0.094], Standard Error of Mean 0.0305

3. Secondary Outcome: Characterize Dose Response of UNR844 as Measured by Change From Baseline in Monocular (Better-seeing Eye) Distance-corrected Near Visual Acuity (DCNVA) at Month 3
Description: Characterize dose response of UNR844 as measured by change from baseline at Month 3 in monocular (better-seeing eye) DCNVA in Logarithm of Minimum Angle of Resolution (logMAR), at 40cm. A low logMAR score represents good vision while a high logMAR score represents bad vision.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: logMAR
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
logMAR | -0.056 (0.0194) | -0.075 (0.0198) | -0.081 (0.0210) | -0.059 (0.0194) | -0.085 (0.0206)
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.284, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.029, 95% CI 2-sided [-0.024 to 0.083], Standard Error of Mean 0.0273
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.711, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.010, 95% CI 2-sided [-0.044 to 0.065], Standard Error of Mean 0.0278
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.871, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.005, 95% CI 2-sided [-0.051 to 0.060], Standard Error of Mean 0.0284
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Mixed-effect Model for Repeated Measures model-based two-sided t-test; p = 0.329, Mixed-effect Model for Repeated Measures; Least Squares Mean = 0.027, 95% CI 2-sided [-0.027 to 0.080], Standard Error of Mean 0.0273

4. Secondary Outcome: Percentage of Participants Gaining at Least 0.30 logMAR in Binocular Distance-corrected Near Visual Acuity (DCNVA) (Without Near Correction) From Baseline at Month 3
Description: Percentage of participants gaining at least 0.3 logMAR in binocular DCNVA compared to baseline at Month 3. DCNVA is measured in Logarithm of Minimum Angle of Resolution (logMAR) at 40 cm, with subjects corrected for any distance refraction error. A low logMAR score represents good vision while a high logMAR score represents bad vision.
  Percentages were derived from Rubin's rule by integrating all results from multiple imputations. For subjects with missing DCNVA at Month 3, the value of DCNVA was imputed and dichotomized to derive the endpoint of gaining of 3 lines.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
Percentage of participants | 4.4 [0.00 to 10.30] | 9.3 [0.78 to 17.90] | 14.9 [3.89 to 25.92] | 5.1 [0.00 to 11.70] | 4.6 [0.00 to 10.72]
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.516, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.95, 95% CI 2-sided [0.083 to 10.847]
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.177, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 2.45, 95% CI 2-sided [0.367 to 16.398]
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.079, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 3.65, 95% CI 2-sided [0.604 to 22.094]
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.476, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 1.07, 95% CI 2-sided [0.136 to 8.381]

5. Secondary Outcome: Percentage of Participants Gaining at Least 0.30 logMAR in Monocular (Worse-seeing Eye) Distance-corrected Near Visual Acuity (DCNVA) (Without Near Correction) From Baseline at Month 3
Description: Percentage of participants gaining at least 0.3 logMAR in monocular (worse-seeing eye) DCNVA compared to baseline at Month 3. DCNVA is measured in Logarithm of Minimum Angle of Resolution (logMAR) at 40 cm, with subjects corrected for any distance refraction error. A low logMAR score represents good vision while a high logMAR score represents bad vision.
  Percentages were derived from Rubin's rule by integrating all results from multiple imputations. For subjects with missing DCNVA at Month 3, the value of DCNVA was imputed and dichotomized to derive the endpoint of gaining of 3 lines.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
Percentage of participants | 13.0 [3.32 to 22.62] | 9.0 [0.61 to 17.33] | 8.7 [0.00 to 17.82] | 10.0 [1.31 to 18.62] | 11.9 [2.16 to 21.71]
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.577, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.201 to 3.726]
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.804, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.52, 95% CI 2-sided [0.113 to 2.353]
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.850, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.34, 95% CI 2-sided [0.045 to 2.602]
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.684, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.157 to 3.080]

6. Secondary Outcome: Percentage of Participants Gaining at Least 0.30 logMAR in Monocular (Better-seeing Eye) Distance-corrected Near Visual Acuity (DCNVA) (Without Near Correction) From Baseline at Month 3
Description: Percentage of participants gaining at least 0.3 logMAR in monocular (better-seeing eye) DCNVA compared to baseline at Month 3. DCNVA is measured in Logarithm of Minimum Angle of Resolution (logMAR) at 40 cm, with subjects corrected for any distance refraction error. A low logMAR score represents good vision while a high logMAR score represents bad vision.
  Percentages were derived from Rubin's rule by integrating all results from multiple imputations. For subjects with missing DCNVA at Month 3, the value of DCNVA was imputed and dichotomized to derive the endpoint of gaining of 3 lines.
Time Frame: Baseline, Month 3
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
Percentage of participants | 6.3 [0.00 to 13.20] | 9.4 [0.77 to 17.93] | 0.3 [0.00 to 2.50] | 2.8 [0.00 to 7.88] | 7.8 [0.00 to 16.13]
Statistical Analysis 1: Comparison: UNR844 5 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.728, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.56, 95% CI 2-sided [0.089 to 3.593]
Statistical Analysis 2: Comparison: UNR844 13.3 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.428, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.242 to 5.529]
Statistical Analysis 3: Comparison: UNR844 23 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.500, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.00, 95% CI 2-sided [lower limit 0.000] (NA when n = 1.)
Statistical Analysis 4: Comparison: UNR844 30 mg/mL vs Placebo Ophthalmic Solution; Test type: Other — Logistic model-based one-sided t-test; p = 0.851, Multiple Imputation, Logistic Regression; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.026 to 3.070]

7. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths were collected from first dose of study medication to 30 days after the last dose of study medication, for a maximum timeframe of approx. 4 months.
  Post-treatment deaths were collected from day 31 after last dose of study medication to end of study, up to approx. 1 year and 1 month.
  All deaths refer to the sum of on-treatment and post-treatment deaths.
Time Frame: On-treatment: up to 121 days, approx. 4 months. Off treatment: up to approx. 1 year and 1 month
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo Ophthalmic Solution
Number analyzed (Participants) | 48 | 48 | 44 | 48 | 46
Participants
  Total Deaths | 0 | 0 | 0 | 0 | 1
  On-Treatment Deaths | 0 | 0 | 0 | 0 | 0
  Post-Treatment Deaths | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment (Max treatment exposure = 115 days) plus a maximum of 9 months post treatment, up to a maximum duration of approx. 1 year and 1 month.
Groups:
- Placebo: Placebo ophthalmic solution; one drop twice-a-day for three months
- Total: Total
Arm/Group | UNR844 5 mg/mL | UNR844 13.3 mg/mL | UNR844 23 mg/mL | UNR844 30 mg/mL | Placebo | Total
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/44 | 0/48 | 1/46 | 1/234
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/48 | 0/44 | 1/48 | 3/46 | 5/234
Other Adverse Events (participants affected / at risk) | 26/48 | 22/48 | 16/44 | 23/48 | 21/46 | 108/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UNR844 5 mg/mL (N=48) | UNR844 13.3 mg/mL (N=48) | UNR844 23 mg/mL (N=44) | UNR844 30 mg/mL (N=48) | Placebo (N=46) | Total (N=234)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1
Pancreatic cystadenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Myelitis transverse (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UNR844 5 mg/mL (N=48) | UNR844 13.3 mg/mL (N=48) | UNR844 23 mg/mL (N=44) | UNR844 30 mg/mL (N=48) | Placebo (N=46) | Total (N=234)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1
Asthenopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Blepharitis (Eye disorders) | 0 | 1 | 1 | 1 | 2 | 5
Central serous chorioretinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 3 | 0 | 1 | 4
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 2
Corneal epithelium defect (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 1 | 1 | 1 | 0 | 3
Episcleritis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Erythema of eyelid (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Eye pain (Eye disorders) | 0 | 1 | 1 | 0 | 1 | 3
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 2
Eyelid cyst (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eyelid rash (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Eyelid skin dryness (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Narrow anterior chamber angle (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Noninfective conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Punctate keratitis (Eye disorders) | 1 | 0 | 0 | 2 | 0 | 3
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 1 | 3
Injection site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 2 | 1 | 7
Sensation of foreign body (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 1 | 2 | 4
COVID-19 (Infections and infestations) | 15 | 10 | 5 | 8 | 8 | 46
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 3 | 2 | 0 | 0 | 6
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Peritonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Rocky mountain spotted fever (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 2 | 1 | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 3
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 1 | 3
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 2
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Hormone level abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 2
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Blepharal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1
Bell's palsy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 3
Headache (Nervous system disorders) | 1 | 4 | 2 | 1 | 1 | 9
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Spinal meningeal cyst (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0 | 0 | 2
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Abnormal uterine bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 4
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Menopause (Social circumstances) | 0 | 1 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/03/NCT04806503/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT04806503/SAP_001.pdf